CLINICAL TRIAL: NCT00002270
Title: A Pilot Study of the Efficacy of Recombinant Alpha Interferon (IFN-A2b) and Zidovudine (AZT) in the Treatment of Progressive Multifocal Leukoencephalopathy (PML) Complicating HIV-1 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 074A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-03

CONDITIONS: HIV Infections; Leukoencephalopathy, Progressive Multifocal
Keywords: Leukoencephalopathy, Progressive Multifocal; Interferon Alfa-2b; Drug Evaluation; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Leukoencephalopathy, Progressive Multifocal; Acquired Immunodeficiency Syndrome | interventions — Interferon alpha-2; Zidovudine

INTERVENTIONS:
Drug: Interferon alfa-2b
Drug: Zidovudine

SUMMARY:
To study the effectiveness of alpha interferon (IFN-A2b) and zidovudine (AZT) in treating progressive multifocal leukoencephalopathy (PML) as a complication of HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity by both ELISA and Western blot.
* Biopsy proven progressive multifocal leukoencephalopathy (PML).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Intolerant to interferon.
* Prior or concomitant central nervous system disease (CNS) such as toxoplasmosis, multiple sclerosis (MS), or neurosyphilis.

Patients with the following are excluded:

* Intolerant to interferon.
* Prior or concomitant central nervous system disease (CNS) such as toxoplasmosis, multiple sclerosis (MS), or neurosyphilis.

Prior Medication:

Excluded:

* Patients receiving interferon for other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Miami School of Medicine, Miami, Florida, United States